CLINICAL TRIAL: NCT05148143
Title: Raltitrexed Combined With Oxaplatin as Second Line Treatment for Advanced Malignant Biliary System Tumor
Brief Title: RALOX as Second Line Treatment for Advanced Malignant Biliary System Tumor
Acronym: RALOXBTC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RALOX 202102
Record Dates: First submitted 2021-11-18; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-08

CONDITIONS: Cholangioadenoma
Keywords: cholangioadenoma; first line treatment failure; raltitrexed;; oxaliplatin
MeSH Terms: conditions — Adenoma, Bile Duct

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RALOX (Experimental): Raltitrexed combined with oxaplatin
  Interventions: Drug: Raltitrexed combined with oxaplatin

INTERVENTIONS:
Drug: Raltitrexed combined with oxaplatin — Raltitrexed combined with oxaplatin as second line treatment of cholangiocarcinoma
  Other Names: Sai Wei Jian

SUMMARY:
The purpose of this study was to explore the safety and efficacy of raltitrexed combined with oxaplatin as second line treatment for advanced malignant biliary system tumor.

DETAILED DESCRIPTION:
The purpose of this study was to explore the safety and efficacy of raltitrexed combined with oxaplatin as second line treatment for advanced malignant biliary system tumor. Single arm，phase II study for patients with cholangiocarcinoma or gallbladder carcinoma after first line treatment failure to explore effection and safety of raltitrexed combined with oxaplatin as second line treatment；Sample size：50.

ELIGIBILITY:
Inclusion Criteria

1. 18-75 years old.
2. Patients with unresectable advanced advanced Gallbladder carcinoma or Cholangiocarcinoma confirmed by histology or cytology.
3. First-line chemotherapy failure (toxic side effects can not be tolerated, disease progression during treatment or relapse after treatment) ;Or the disease recurred within 6 months after completion of adjuvant chemotherapy.
4. At least one measurable lesion according to RECIST1.1 criteria.
5. ECOG: 0 ~ 1.
6. Life expectancy ≥ 12 Weeks.
7. The major organs were functioning normally, and the laboratory examination results within 1 week met the following conditions before enrollment:①Absolute neutrophil count (ANC)≥1.5×109/L ②Platelet count（PLT）≥80.0 × 109/L ③Hemoglobin concentration（HB） ≥90g/L④ Total bilirubin（TB）≤1.5×ULN ⑤ Serum creatinine （Cr）≤l.5×ULN ，Endogenous creatinine clearance >60ml/min（Cockcroft-Gault Formula ）⑥Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase(AP): ≤3 ×ULN (≤5 ×ULN for metastases to liver).
8. Sign the informed consent voluntarily.

Exclusion Criteria

1. Allergic to any research drug and its excipients.
2. Prior use of raltitrexed or oxaliplatin.
3. History of other malignancies, except cured Basal cell or squamous Cell Carcinoma of the skin and carcinoma in situ of the cervix.
4. There is a history of brain metastases.
5. History of psychotropic drug abuse and cannot quit or has a mental disorder.
6. Uncontrolled chronic infectious and non-infectious diseases.
7. Active or clinically poorly controlled severe infection
8. Other conditions that the researchers think should be ruled out.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS（Progression Free Survival） | 24 months
  PFS is defined as the time interval from initiation of treatment to the first date of documented tumor progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
ORR | 24 months
  Overall Response Rate
OS | 36 months
  Overall Survival
DCR | 24 months
  Disease Control Rate
Qol ( quality of life ) | 24 months
  EORTC-QLQ-C30 is a cancer-specific instrument
AE | 12 months
  Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Ph.D&MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China